CLINICAL TRIAL: NCT04012047
Title: Headache Inducing Effect of Levcromakalim in Migraine With Aura Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Mohammad Al-Mahdi Al-Karagholi, MD, PhD student, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: Journal-nr.: H-19023571
Record Dates: First submitted 2019-07-04; First posted 2019-07-09 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Headache; Migraine; Aura
Keywords: Levcromakalim
MeSH Terms: conditions — Headache; Migraine Disorders; Epilepsy | interventions — Cromakalim; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levcromakalim (Active Comparator)
  Interventions: Drug: Levcromakalim
- Saline (Placebo Comparator)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Levcromakalim — To investigate the role of levcromakalim compared with placebo in migraine with aura patients
  Arms: Levcromakalim
Drug: Saline — To investigate the role of levcromakalim compared with placebo in migraine with aura patients
  Arms: Saline

SUMMARY:
To investigate the role of KATP channels in migraine with aura patients.

ELIGIBILITY:
Inclusion Criteria:

* Migraine with aura patients of both sexes.
* 18-60 years.
* 50-100 kg.

Exclusion Criteria:

* Headache less than 48 hours before the tests start
* Daily consumption of drugs of any kind other than oral contraceptives
* Pregnant or nursing women.
* Cardiovascular disease of any kind, including cerebrovascular diseases.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2019-07-09 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
Headache | Before (-10 min) and after infusion (+12 hours) of levcromakalim compared with before and after infusion of saline
  Occurrence of headache
Migraine | Before (-10 min) and after infusion (+12 hours) of levcromakalim compared with before and after infusion of saline
  Occurrence of migraine
Aura | Before (-10 min) and after infusion (+12 hours) of levcromakalim compared with before and after infusion of saline
  Occurrence of aura

SECONDARY OUTCOMES:
The area under the curve (AUC) for headache | Before (-10 min) and after infusion (+12 hours) of levcromakalim compared with before and after infusion of saline
  Headache intensity
Family history | After including the patients in the study.
  Direct interview with the 1 st degree family memeber for included patients according to international classification of headaches.
Heart rate | Before (-10 min) and after infusion (+2 hours) of levcromakalim compared with before and after infusion of saline
  Change in heart rate measured in Beats per minute (BPM)
Blood pressure | Before (-10 min) and after infusion (+2 hours) of levcromakalim compared with before and after infusion of saline
  Change in blood pressure measured in mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Messoud Ashina, Study Director — Danish Headache Center
Locations (1):
- Danish headache center, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Al-Karagholi MA, Ghanizada H, Nielsen CAW, Hougaard A, Ashina M. Opening of ATP sensitive potassium channels causes migraine attacks with aura. Brain. 2021 Sep 4;144(8):2322-2332. doi: 10.1093/brain/awab136. PMID 33768245